CLINICAL TRIAL: NCT06193616
Title: Evaluating Baseline Predictors Including Total Kidney Volume, of Chronic GFR Decline and Other Clinical Outcomes in Outpatients With ADPKD and Stage IV CKD on Chronic Treatment With Octreotide LAR: a Retrospective, Observational Study
Brief Title: Outcome of ADPKD With Octreotide LAR
Acronym: ADPKD648
Status: Active, not recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: ADPKD648
Record Dates: First submitted 2023-12-14; First posted 2024-01-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Autosomal Dominant Polycystic Kidney
Keywords: ADPKD; Total kidney volume; Octreotide; Sandostatina LAR
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Octreotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Octreotide — All consenting patients treated with octreotide LAR according to Determina AIFA n. 1264 del 3 August 2018 and fulfilling the selection criteria will be collected at prespecified time-points according to the routine visits scheduled for these patients and the periodic follow-up visits till dialysis initiation as described in the AIFA indication on GU Serie Generale n.5 del 08-01-2020.
  Other Names: Octreotide LAR

SUMMARY:
In this observational, retrospective study we will primarily aim at evaluating the independent role of baseline clinical and laboratory parameters, including TKV, in the prediction of long term chronic GFR decline and other clinical outcomes and, secondarily, the relationships between GFR and TKV changes over time, in a cohort of ADPKD patients with Stage IV CKD on chronic treatment with octreotide LAR and routinely monitored with serial GFR, TKV and clinical evaluations, at the outpatient clinic of the Nephrology Unit of the Azienda Socio-Sanitaria Territoriale Papa Giovanni XXIII, Bergamo, Italy.

DETAILED DESCRIPTION:
Autosomal Dominant Polycystic Kidney Disease (ADPKD), the most common hereditary cystic renal disease, has an incidence of 1 in 800 live births and accounts for 7-10% of patients on dialysis in developed countries. ADPKD shows genetic heterogeneity, with two main genes implicated, namely the PKD gene 1 (85%-90% of the cases) and the PKD gene 2 (10-15% of the cases) which encode for proteins policystin 1 and policystin 2, respectively. Clinically, ADPKD is characterized by renal and extra renal manifestations. In the kidneys, multiple cysts grow from distal and collecting tubular epithelial cells producing progressive renal enlargement with initially relatively stable renal function. Thereafter, both tubular and secondary interstitial damage lead to faster renal loss and end-stage renal disease (ESRD) in approximately half of the patients affected in their fifth or sixth decade of life. More than 50% of the patients display hepatic cysts generated from cholangiocytes proliferation and fluid secretion as well as other extra-renal manifestations such as pancreatic and intestinal cysts, increased risk of aortic aneurysms, heart-valve defects and sudden death due to rupture of intracerebral aneurysms. The precise molecular pathogenic mechanisms of ADPKD are not completely understood, but experimental models in renal tubular cells suggest that defect in policystin 1 or policystin 2 carry out to decrease intracellular calcium and increase cAMP (Cyclic adenosine monophosphate) levels changing the cell toward a proliferative and secretor phenotype. Cysts growth and enlargement are mainly consequence of epithelial cell proliferation and fluid chloride secretion through apical channels dependent of cAMP. Likewise, for hepatic cyst development, the proposed mechanisms are linked to abnormalities in epithelial cell proliferation and secretion in response to high intracellular cAMP concentrations secondary to policystin defects.

Since the proliferative and secretory phenotype of renal and hepatic cells appear to be supported by an increase in intracellular levels of cAMP, it has been hypothesized that interventions able to reduce cAMP synthesis or accelerate the metabolism could have a protective effect against disease progression in ADPKD patients. With this rationale, some clinical studies have aimed to test the effect of drugs capable of reducing the bioavailability of intracellular cAMP like somatostatin analogues such as octreotide, lanreotide, pasireotide and others. Moreover, antidiuretic hormone receptor antagonists, such as Tolvaptan act on the same mechanism. On the basis of the results of these clinical trials, Tolvaptan has been approved by international regulatory authorities to slow the progression of cyst development and renal failure associated with ADPKD in adults with stage 1 to 3 CKD (chronic kidney disease), with evidence of rapidly progressing disease. However, major limitation to the use of Tolvaptan in clinical practice exist due to serious liver toxicity and the polyuric effect that has a major impact on treatment tolerability and patient adherence to therapy.

In recent years, ALADIN and ALADIN 2 studies coordinated by researchers from the Istituto di Ricerche Farmacologiche Mario Negri IRCCS with the collaboration of nephrologists from several Italian Nephrology Units, have shown that the somatostatin analogue octreotide Long Acting Release (LAR) has major nephroprotective effects in patients with ADPKD. ALADIN clinical study showed that a 3-year treatment with octreotide LAR significantly slowed kidney volume growth and disease progression in adult ADPKD patients with preserved or moderately impaired renal function(13). More recently, the ALADIN 2 clinical trial found that octreotide LAR slows kidney volume growth and progression to the combined endpoint of doubling of serum creatinine or end stage renal disease (ESRD) in ADPKD patients with advanced CKD (stages 3b to 4). In the latter study, the protective effect of octreotide LAR against progression to ESRD was fully driven by nephroprotection in ADPKD patients with CKD stage 4. These findings suggested that even in later pre-terminal stages of ADPKD, when the kidney architecture is largely disrupted, octreotide LAR may still exert a specific and clinically relevant protective effect against the progression to ESRD. On the basis of the results of the ALADIN 2 study, published in the PLOS Medicine journal, in August 2018, the Italian Medicines Agency (AIFA), has included octreotide LAR (Determina n. 1264 of 3 August, 2018 and subsequent amendments) in the list of prescription drugs according to the provisions of Law 648/96 for patients with ADPKD and severe renal insufficiency (stage 4: estimated glomerular filtration rate [eGFR] 30-15 ml/min/1.73 m2 measured by the MDRD 4-variable equation). Actually, in Italy, only a minority of Nephrologists have started to use octreotide LAR for the treatment of ADPKD patients in every day clinical practice, partly due to theoretical considerations, but also as a result of administrative obstacles to its prescription as well as practical difficulties in treatment administration. Thus, a substantial proportion of ADPKD patients is left without this effective treatment.

Total kidney volume (TKV) increase is acknowledged by the scientific community to be the dominant feature of ADPKD progression. Moreover, baseline TKV was found to predict GFR decline over time. TKV can also serve as an indicator to evaluate the efficacy of candidate therapeutic agents that target cyst formation and growth in ADPKD patients. Clinical studies have highlighted that drug treatment in these patients could limit kidney enlargement earlier and to a greater extent than slowing renal function decline. Finally, TKV has been recently recognized by the EU and US regulatory agencies as an enrichment biomarker and a possible surrogate endpoint. In response to a request from the FDA, the Polycystic Kidney Disease Outcomes Consortium (PKDOC) gathered TKV data from more than 2 thousand patients with ADPKD to track the decline in eGFR as a function of baseline TKV. As a result of the PKDOC findings, in 2015, the US Food and Drug Administration (FDA) published a letter of support, and the European Medicines Agency (EMA) a positive qualification opinion for TKV as an exploratory prognostic biomarker for enrichment in ADPKD clinical trials. In 2016, the FDA qualified TKV as a prognostic biomarker and in 2018 it further designated TKV as a reasonably likely surrogate endpoint.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD patients with criteria for the prescription of octreotide LAR according to Law n. 648, 23 December 1996: ≥ 18 year-old; Clinical and instrumental diagnosis of ADPKD; Estimated GFR (MDRD): ≥ 15 ml/min/1.73m2 and <30 ml/min/1.73m2.
* Written informed consent to participate in the observational study and to the use of recorded data for research purposes.
* Availability of an adequate (for quantitative volumetric analyses) non-contrast enhanced Computed Tomography (CT) scan acquired before starting octreotide-LAR therapy.
* Follow-up of at least six months (eg. up to the first post-treatment GFR evaluation from the start of chronic octreotide LAR treatment).

Exclusion Criteria:

* Legal incapacity or limited legal capacity.
* Contraindications to the prescription of octreotide LAR according to Law n. 648, 23 December 1996.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ADPKD who have undergone chronic treatment with octreotide LAR (in accordance with Law N. 648 of December23, 1996), suffering from stage IV CKD and who have been regularly followed, through serial measurements of GFR and TKV and clinical examinations, at the outpatient clinic of the Nephrology Unit at the ASST Papa Giovanni XXIII in Bergamo, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
GFR change over time | change from start (day 0) and month 6,12,18,24,30,36,42,48
  Assessed by six-monthly routine iohexol plasma clearance and annual TKV measurements

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- ASST HPG23 - Unità di Nefrologia, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caroli A, Perico N, Perna A, Antiga L, Brambilla P, Pisani A, Visciano B, Imbriaco M, Messa P, Cerutti R, Dugo M, Cancian L, Buongiorno E, De Pascalis A, Gaspari F, Carrara F, Rubis N, Prandini S, Remuzzi A, Remuzzi G, Ruggenenti P; ALADIN study group. Effect of longacting somatostatin analogue on kidney and cyst growth in autosomal dominant polycystic kidney disease (ALADIN): a randomised, placebo-controlled, multicentre trial. Lancet. 2013 Nov 2;382(9903):1485-95. doi: 10.1016/S0140-6736(13)61407-5. Epub 2013 Aug 21. PMID 23972263
- [Background] Perico N, Ruggenenti P, Perna A, Caroli A, Trillini M, Sironi S, Pisani A, Riccio E, Imbriaco M, Dugo M, Morana G, Granata A, Figuera M, Gaspari F, Carrara F, Rubis N, Villa A, Gamba S, Prandini S, Cortinovis M, Remuzzi A, Remuzzi G; ALADIN 2 Study Group. Octreotide-LAR in later-stage autosomal dominant polycystic kidney disease (ALADIN 2): A randomized, double-blind, placebo-controlled, multicenter trial. PLoS Med. 2019 Apr 5;16(4):e1002777. doi: 10.1371/journal.pmed.1002777. eCollection 2019 Apr. PMID 30951521
- [Background] Trillini M, Caroli A, Perico N, Remuzzi A, Brambilla P, Villa G, Perna A, Peracchi T, Rubis N, Martinetti D, Caruso M, Leone VF, Cugini D, Carrara F, Remuzzi G, Ruggenenti P; TOOL Study Group. Effects of Octreotide-Long-Acting Release Added-on Tolvaptan in Patients with Autosomal Dominant Polycystic Kidney Disease: Pilot, Randomized, Placebo-Controlled, Cross-Over Trial. Clin J Am Soc Nephrol. 2023 Feb 1;18(2):223-233. doi: 10.2215/CJN.0000000000000049. PMID 36754009